CLINICAL TRIAL: NCT03860350
Title: Aged Garlic Extract (Kyolic) Study at Lund University, Sweden
Brief Title: Aged Garlic Extract Study
Acronym: AGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Sandra Lindstedt Ingemansson, Senior Consultant and Associate Professor, Lund University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: DNR2016/745
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Coronary Artery Disease; Microcirculation; Biomarkers
Keywords: garlic
MeSH Terms: conditions — Coronary Artery Disease | interventions — kyolic

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled prospective study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aged Garlic Extract (Active Comparator): The participants will ingest 600 mg of Aged Garlic Extract in two capsules two times a day i.e. 1200 mg/day during a period of one year.
  Interventions: Dietary Supplement: Aged Garlic Extract
- Placebo (Placebo Comparator): The participants will ingest 600 mg of placebo in two capsules two times a day i.e. 1200 mg/day during a period of one year.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Aged Garlic Extract
  Other Names: Kyolic
  Arms: Aged Garlic Extract
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The primary intention of the study is to examine the effect of aged garlic extract (AGE) on the absolute change in coronary artery calcium (CAC). The second intention is to examine the effect of AGE on inflammatory biomarkers and microcirculation. It is a double blind placebo controlled study. The participants will ingest AGE during a period of one year. The CAC will be controlled by computer tomography (CT) scan; the inflammatory biomarkers through blood sample test and the microcirculation through laser speckel imagining and laser doppler before and after the one year period of AGE ingestion.

DETAILED DESCRIPTION:
Objectives:

Effect on coronary artery atherosclerosis / the progression of atherosclerosis Effect on inflammatory and oxidation biomarkers Cholesterol lowering effect Effect on microcirculation

Type of study:

Randomized double blind controlled trial

Number of patients: 80 patients

Duration of the study:

The patients will be studied for one year after they have entered the study. The total time of the study duration from the including date of the first patient to the analysis of the last patient entering the study estimated to be 2-3 years. An inclusion rate off 1 to 2 patients per week.

Treatment:

Dose: Treated with a placebo capsule or a capsule containing a total of AGE 2400 mg daily for 1 year (2 Kyolic capsule (600 mg) twice daily).

Methods:

Placebo-controlled double blind randomized trial to determine whether AGE can influence the rate of atherosclerosis plaque burden measured by coronary artery calcium, improve vascular function and microcirculation and favorably change biomarkers of oxidative stress.

Randomization:

The participants are assigned to AGE or placebo in a double-blinded manner, using numbered containers assigned to a computer-generated randomization chart by a nurse coordinator.

ELIGIBILITY:
Inclusion Criteria:

* CAC score >10
* Framingham risk score (10 % or above)
* Subjects are required to be on stable concomitant medications for at least 12 weeks prior to randomization
* Subjects with diabetic must have HbA1C < 8.0, and stable HbA1C level variation range within 0.5% for three months.

Exclusion Criteria:

* Hypersensitivity to AGE therapy,
* Unstable medical, psychiatric, or substance abuse disorder that may interfere with continuation in the study,
* Weight ≥325 pounds,
* Bleeding disorder,
* History of myocardial infarction,
* Stroke
* Life-threatening arrhythmia within prior 6 months,
* Resting hypotension (systolic < 90 mmHg) or hypertension (resting blood pressure >170/110)
* Heart failure NYHA class III or IV,
* History of malignancy within the last 5 years (other than skin cancer) or evidence of active cancer which would require concomitant cancer chemotherapy
* Serum creatinine >1.4 mg/dl
* Triglycerides > 400 at baseline visit
* Diabetic subjects with HbA1C > 8 %,
* Drug or alcohol abuse
* Conditions interfering with accurate assessment of coronary calcification (metal clips, bypass patients, intracoronary stents) and drug absorption (partial ileal bypass or malabsorption syndrome).
* Current use of anticoagulants (except for antiplatelet agents)
* Chronic renal failure
* Liver failure
* Hematological or biochemical values at baseline visit outside the reference ranges considered as clinically significant.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in coronary artery calcium (CAC) score | One year
  CAC is to be defined as a plaque of at least three contiguous pixels (area 1.02 mm 2) with a density of > 130 Hounsfield units. The lesion score are to be calculated by multiplying the lesion area by a density factor derived from the maximal Hounsfield unit within this area, as described by Agatston S, Janowitz WR, Hildner FJ et al. Quantification of coronary artery calcium using ultrafast computed tomography. J Am Coll Cardiol 1990; 15: 827-832. CAC score is measured at baseline and after one year follow-up and the difference is calculated.

SECONDARY OUTCOMES:
The changes in inflammatory biomarkers. | One Year
  Changes in C-reactive protein (CRP mg/L)
The changes in Interleukin-6 (IL-6) | One Year
  Changes in IL-6 (ng/L)
The changes in inflammatory biomarkers. | One Year
  Changes in Homocystein (µmol/L)
The changes in the microcirculation measured by Laser Doppler velocimetry | One Year
  Laser Doppler Flowmetry (LDF) is a non-invasive method to estimate the blood perfusion in the microcirculation. The advantage of the technique is that LDF provide a continuous or near continuous record of the microvascular blood flow. No current laser Doppler instrument can present absolute perfusion values (e.g. ml/min/100 gram tissue). Measurements are expressed as perfusion units (PU) which are arbitrary. The changes in PU will be measured.
Changes in Low Density Lipoprotein | One Year
  Changes of Low Density Lipoprotein (LDL) mmol/L
Changes in Triglycerides | One Year
  Changes of Triglycerides mmol/L.
Changes in Cholesterol | One Year
  Changes of cholesterol mmol/L.
Changes in High Density Lipoprotein | One Year
  Changes of High Density Lipoprotein(HDL) mmol/L,
Changes in lipid profile | One Year
  Apolipoprotein B (mmol/L)/Apolipoprotein A1 (mmol/L)
Changes in blood sugar | One Year
  Changes in fastening blood glucose measured as mmol/L
Changes in Blood pressure | One Year
  Changes of blood pressure Systolic and Diastolic presented as mmHg.
Changes in BMI | One Year
  Changes in BMI measured as weight (kg) and height (m) and will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Lindstedt, MD, PhD, Principal Investigator — Skane University Hospital
Locations (1):
- Skane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agatston AS, Janowitz WR, Hildner FJ, Zusmer NR, Viamonte M Jr, Detrano R. Quantification of coronary artery calcium using ultrafast computed tomography. J Am Coll Cardiol. 1990 Mar 15;15(4):827-32. doi: 10.1016/0735-1097(90)90282-t. PMID 2407762
- [Background] Lindstedt S, Malmsjo M, Hansson J, Hlebowicz J, Ingemansson R. Microvascular blood flow changes in the small intestinal wall during conventional negative pressure wound therapy and negative pressure wound therapy using a protective disc over the intestines in laparostomy. Ann Surg. 2012 Jan;255(1):171-5. doi: 10.1097/SLA.0b013e31823c9ffa. PMID 22104565
- [Background] Lindstedt S, Malmsjo M, Hlebowicz J, Ingemansson R. Comparative study of the microvascular blood flow in the intestinal wall, wound contraction and fluid evacuation during negative pressure wound therapy in laparostomy using the V.A.C. abdominal dressing and the ABThera open abdomen negative pressure therapy system. Int Wound J. 2015 Feb;12(1):83-8. doi: 10.1111/iwj.12056. Epub 2013 Mar 21. PMID 23517436
- [Background] Lindstedt S, Malmsjo M, Ingemansson R. No hypoperfusion is produced in the epicardium during application of myocardial topical negative pressure in a porcine model. J Cardiothorac Surg. 2007 Dec 6;2:53. doi: 10.1186/1749-8090-2-53. PMID 18062803
- [Background] Lindstedt S, Malmsjo M, Ingemansson R. Blood flow changes in normal and ischemic myocardium during topically applied negative pressure. Ann Thorac Surg. 2007 Aug;84(2):568-73. doi: 10.1016/j.athoracsur.2007.02.066. PMID 17643636
- [Background] Budoff MJ, Ahmadi N, Gul KM, Liu ST, Flores FR, Tiano J, Takasu J, Miller E, Tsimikas S. Aged garlic extract supplemented with B vitamins, folic acid and L-arginine retards the progression of subclinical atherosclerosis: a randomized clinical trial. Prev Med. 2009 Aug-Sep;49(2-3):101-7. doi: 10.1016/j.ypmed.2009.06.018. Epub 2009 Jun 30. PMID 19573556
- [Derived] Wlosinska M, Nilsson AC, Hlebowicz J, Fakhro M, Malmsjo M, Lindstedt S. Aged Garlic Extract Reduces IL-6: A Double-Blind Placebo-Controlled Trial in Females with a Low Risk of Cardiovascular Disease. Evid Based Complement Alternat Med. 2021 Mar 31;2021:6636875. doi: 10.1155/2021/6636875. eCollection 2021. PMID 33868439
- [Derived] Wlosinska M, Nilsson AC, Hlebowicz J, Hauggaard A, Kjellin M, Fakhro M, Lindstedt S. The effect of aged garlic extract on the atherosclerotic process - a randomized double-blind placebo-controlled trial. BMC Complement Med Ther. 2020 Apr 29;20(1):132. doi: 10.1186/s12906-020-02932-5. PMID 32349742